CLINICAL TRIAL: NCT06123611
Title: Pediatric Trauma Centers RE-AIM at Gun Safety - Adopting Comprehensive Training for FireArm Safety in Trauma Centers
Brief Title: Pediatric Trauma Centers RE-AIM at Gun Safety
Acronym: ACTFAST
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Children's Hospitals and Clinics of Minnesota (Other); University of Utah (Other); Rhode Island Hospital (Other); Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00407213; CE003620 (Other Grant/Funding Number: Centers for Disease Control and Prevention)
Record Dates: First submitted 2023-11-01; First posted 2023-11-09 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Firearm Injury; Safety Issues
MeSH Terms: interventions — Trauma Centers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): In the pre-implementation period, all trauma patients will receive standard routine care. Which may include some screening and counseling on gun safety.
- ACTFAST Intervention (Experimental): During the implementation and maintenance periods, all trauma patients will receive study activities including firearm access screening, counseling on safe storage practices, and referral to safe storage and other community resources as appropriate.
  Interventions: Behavioral: Adopting Comprehensive Training for FireArm Safety in Trauma centers

INTERVENTIONS:
Behavioral: Adopting Comprehensive Training for FireArm Safety in Trauma centers — Firearm access screening, brief firearm safe storage intervention, and referral to community and preventive health resources
  Arms: ACTFAST Intervention

SUMMARY:
Universal firearm injury and violence prevention counseling of parents and patients has been recommended by multiple national organizations for over a decade, yet clinicians rarely deliver this counseling. Barriers to its implementation must be addressed in order to effectively deliver firearm related injury prevention efforts. This study will implement a universal firearm injury prevention initiative within a national cohort of three pediatric trauma centers. The investigator's long-term goal is to demonstrate best practices for pediatric trauma center-based firearm injury prevention strategies that promote safe storage practices and reduce firearm related injury and death. This research will test the effectiveness of a comprehensive training strategy for improving the implementation of a universal firearm injury prevention effort, ACTFAST (Adopting Comprehensive Training for FireArm Safety in Trauma centers), to 1) increase the adoption, implementation and sustainability of a universal firearm injury prevention initiative within participating pediatric level 1 trauma centers; 2) increase firearm safety knowledge, attitudes and safe firearm storage practices among parents of pediatric trauma patients and youth patients treated within participating pediatric level 1 trauma centers, and 3) increase trauma center clinicians' firearm safety knowledge and confidence in delivering a firearm safety intervention.

ELIGIBILITY:
For parents/guardians of pediatric trauma patients:

Inclusion Criteria:

* live with an admitted pediatric trauma patient at a participating trauma center
* be fluent in English or Spanish

Exclusion Criteria:

- family members who do not live with the admitted pediatric trauma patient

For youth trauma patients:

Inclusion Criteria:

* Must be between the ages of 11-17 years
* admitted to a participating trauma inpatient service for an injury
* fluent in English or Spanish
* able to provide written assent and parent able to provide written consent

Exclusion Criteria:

* Youth who are prisoners or in police custody
* Youth who are admitted due to suicide attempt
* Youth with acute conditions that would preclude provision of informed consent (i.e., acute psychosis, altered mental status, cognitive impairment)

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-02-25 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Implementation of Intervention | 3 years
  This outcome will be measured using chart review protocols examining rates of firearm access screening, documentation of firearm safety counseling, documentation of referral to community based resources and connection to medical homes as well as patient hospitalization characteristics including admission diagnosis, injury severity and patient demographic characteristics.
Parent firearm safety attitudes and behaviors | 3 years
  This outcome will be measured using parent survey and interview adapted from prior work by the study team.

SECONDARY OUTCOMES:
Clinician firearm safety knowledge and confidence | 3 years
  This outcome will be measured using clinician surveys derived from multiple sources developed through the prior work of members of the study team.
Adolescent patient firearm safety attitudes and behaviors | 3 years
  Measure firearm injury prevention knowledge, attitudes and safe firearm practices of adolescent trauma patients (11-17 years) within participating pediatric level 1 trauma centers. This outcome will be measured using patient survey and interview adapted from prior work by the study team.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Hoops, MD, PhD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
At the conclusion of the study, deidentified data will be made publicly available. Due to the sensitive nature of the topics being discussed, individual participant data will not be made available to other researchers outside of the study team.